CLINICAL TRIAL: NCT01797510
Title: Mayo-Sessions Clinical Trial
Brief Title: Feasibility Study for a Web Based Health Coaching Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Marc R. Matthews, Assistant Professor, Department of Family Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-008958
Record Dates: First submitted 2013-02-20; First posted 2013-02-22 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching (Experimental): Interventional web based coaching study
  Interventions: Behavioral: Web Based Health Coaching
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Web Based Health Coaching
  Arms: Coaching

SUMMARY:
This study is designed to compare an intensive lifestyle and activity coaching program ("Sessions") to usual care for diabetic patients who are sedentary. The question to be answered is whether the Sessions program improves clinical or patient centric outcomes.

Recruitment is through invitiation only.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients age 18 or greater

Exclusion Criteria:

* Patients aged 17 or less,
* Patients with cognition impaired such that they could not comprehend enrollment materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Biometrics | 6 months
  BMI, Blood Pressure

CONTACTS AND LOCATIONS:
Overall Officials: Marc Matthews, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States